CLINICAL TRIAL: NCT01194011
Title: Study on Nation-wide Health Care Quality Information Openness and Transparency Mechanism Establishment
Status: No longer available | Type: Expanded Access
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Yaw-Tang Shih, Taiwan College of Healthcare Executives
Other Study IDs: 99010
Record Dates: First submitted 2010-06-02; First posted 2010-09-02 (Estimated); Last update posted 2010-09-02 (Estimated); Status verified 2010-06

CONDITIONS: Valuable Suggestions to Improve Health Care Quality Transparent and Accessible Medical Care
Keywords: Health care quality, information openness, health care information website
MeSH Terms: interventions — Surveys and Questionnaires; Quality of Health Care

INTERVENTIONS:
Behavioral: questionnaire — This research tool was a written questionnaire, did not do invasive or the subjects are exposed to physical danger on the experiment, so now there is no harm in this research and test more than minimal risk.
  Other Names: Health care quality, information openness, health care information website

SUMMARY:
Research objectives To provide people with sufficient information regarding health care and to improve its quality, this research endeavors to discuss the establishment of a health care information openness and transparency mechanism within the framework of the National Health Insurance system. This research also evaluates whether the transparency of health care quality information makes care givers provide better quality. Meanwhile, when appropriate information and quality index are presented to patients, patients shall have more knowledge about what they are dealing with, hence less misunderstanding between hospitals and patients would occur.

Research Methods

1. To revise indicators based on international trends, related literature and the need of people.
2. To present 50 sets of quality indicator statistically on the website, and provide updated information about the first 10 sets.
3. To analyze and explain the outcome and purposes of the indicator to the public.
4. To estimate the possible trend for the coming year, and provide adaptive strategy.
5. To promote the website, and hold workshops in all six regions of Taiwan.
6. To make the website linked to the top 5 most populated official and unofficial websites.
7. To respond to questions on the forum of the website daily, and maintain the system, update the website regularly.
8. To complete the acceptability survey on health care institutions and people.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient ; healthy subjects patients

Exclusion Criteria:

* The plan excluded child / children and other minors who were the target respondents, mainly to investigate the medical information for public acceptance of the site, child / children is not suitable, so as to adults as the main investigation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Lan-Chi Tai, Master, Principal Investigator — Taiwan College of Healthcare Executives